CLINICAL TRIAL: NCT03390049
Title: Randomized Controlled Trial of Fractional CO2 Laser vs Sham Laser for Women With Provoked Vestibulodynia Who Have Failed Conservative Management
Brief Title: Randomized CO2 vs Sham Laser Treatment of Provoked Vestibulodynia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00043442
Record Dates: First submitted 2017-12-26; First posted 2018-01-04 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2018-02

CONDITIONS: Vestibulodynia
Keywords: SmartXide 2 V 2 LR; MonaLisa Touch; DEKA; Fractional CO2 Laser; Sham Laser; Vulvodynia; PVD; Provoked vestibulodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Each subject will be assigned a study identification number, and demographic and clinical data will be recorded in REDCAP on de-identified data collection forms. The lead research coordinator will maintain the key linking the identification number to each subject in a locked, password-protected site. A random number generator in REDCAP will then randomly assign each subject to either fractional CO2 laser or sham laser.
  The physician administering the laser sessions will be blinded to treatment arm assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fractional CO2 Laser Treatment (Active Comparator): Fractional CO2 laser will be applied to the entire vestibule, anteriorly to the fourchette, and laterally to the labia majora. This takes approximately 5 minutes to complete. A treatment cycle will consist of three laser sessions separated by 6 weeks +/- 1 week. The procedures will take place in the outpatient clinic. EMLA cream will be applied to the introitus for 20 minutes and wiped clean and dried prior to each laser session. Subjects will be advised to avoid intercourse for at least 3 days after each laser session because a mild inflammatory reaction may last up to 48 hours after a laser session. Topical lidocaine 5% ointment may be used for any vulvar discomfort post-procedure.
  Interventions: Device: Fractional CO2 Laser Treatment
- Sham Laser Treatment (Sham Comparator): A treatment cycle will consist of three laser sessions separated by 6 weeks +/- 1 week. The procedures will take place in the outpatient clinic. Subjects assigned to sham laser will undergo the same pre-treatment with EMLA cream and will receive the same post-treatment instructions as the fractional CO2 laser subjects.
  Interventions: Device: Sham Laser Treatment

INTERVENTIONS:
Device: Fractional CO2 Laser Treatment — After obtaining a negative urine pregnancy test, each subject assigned to the fractional CO2 laser treatment arm will undergo laser sessions with the fractional microablative CO2 laser system (SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy) using the flat vulvar probe with the following settings: dot power 26 Watts, dwell time 1000 μs, dot spacing 1000 μm, and smart stack parameter from 1 to 3. Stack 1 is used at baseline; stack 3 is used 6 and 12 weeks after.
  Other Names: Fractional microablative CO2 laser system
  Arms: Fractional CO2 Laser Treatment
Device: Sham Laser Treatment — After obtaining a negative urine pregnancy test, each subject assigned to the sham laser treatment arm will undergo laser sessions with the fractional microablative CO2 laser system (SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy) using the flat vulvar probe. However, these sham laser sessions will administer no fractional CO2 laser energy. To increase the likelihood that subjects assigned to sham laser remain blinded to treatment arm assignment during the study, MonaLisa Touch will provide a software package with settings that allow for reproduction of the sounds generated during a regular fractional CO2 laser session but using 0 Watts of power.
  Other Names: Fractional microablative CO2 laser system
  Arms: Sham Laser Treatment

SUMMARY:
Vulvodynia is a debilitating chronic vulvar pain lasting at least 3 months without a clear identifiable cause that is challenging to treat effectively. Vulvodynia is a common pain condition: its prevalence is estimated at 7-8% in women between the ages of 18 and 40. Vulvodynia that is provoked and localized to the vestibule (provoked vestibulodynia [PVD]) appears to be the most commonly seen in clinical practice. The current treatment approach for PVD follows a trial-and-error strategy from one intervention to another if symptoms fail to remit. Treatment options include reducing vulvar irritation (e.g., by stopping the use of detergents), topical agents (e.g., lidocaine), oral medications, pelvic floor physical therapy, psychotherapy, locally injectable agents (e.g., botulinum toxin A), and surgery (vestibulectomy). Despite the number of available treatment options, treatment failure is common.

Fractional carbon-dioxide (CO2) laser is a technology widely used in dermatology for the treatment of various skin conditions. It has also been found to be an effective and safe treatment modality for symptoms of the genitourinary syndrome of menopause. A recent pilot study explored the use of fractional CO2 laser for the treatment of vestibulodynia in 37 subjects, 67.6% of which reported that their symptoms were "improved" or "very improved" after 3 fractional CO2 laser sessions. In addition, the subjects reported statistically-significant decreases in vulvar pain and dyspareunia scores. Though the results of this pilot study are promising, it was of small sample size and did not control for the placebo effect. In cases of PVD, the placebo effect has been found to have a significant impact on self-reported outcomes. Sham procedures, when performed correctly, can be ethically administered and can significantly reduce study bias.

The primary aim of this study, therefore, is to assess the difference in vulvar pain intensity scores, at baseline and at 6, 12, 16, and 24 weeks post-randomization, in women with refractory PVD assigned to fractional CO2 laser vs sham laser. This study will provide information about the efficacy of this treatment modality in women with a challenging clinical condition. Hypothesis: Administration of 3 sessions of fractional carbon-dioxide laser to the vulvar vestibule of women with refractory provoked vestibulodynia will result in a clinically-significant greater reduction in vulvar pain intensity scores than placebo (sham laser).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Meets the 2015 terminology for the diagnosis of PVD, either type 1 (chronic vulvar pain since first attempts at intercourse and/or other penetrative activities) or type 2 (chronic vulvar pain with intercourse and/or other penetrative activities following a period of no vulvar pain)
* Vulvar pain is localized to the vestibule and provoked by vaginal intercourse, other penetrative activities (e.g., tampon insertion, self-stimulation) and/or pressure exerted on the vestibule (e.g., due to tight-fitting clothing, cycling)
* Vestibular pain is elicited with cotton-swab test during screening medical examination
* Subject did not experience significant symptom improvement with prior therapy following a minimum of 2 standard-of-care treatments for PVD

Exclusion Criteria:

* Currently receiving any type of treatment for PVD, including topical agents (e.g., lidocaine), oral medications (e.g., tricyclic antidepressants, anticonvulsants), pelvic floor physical therapy, psychotherapy, or locally injectable agents (e.g., botulinum toxin A)
* Generalized vulvar pain
* Unprovoked vulvar pain
* History of vestibulectomy
* Any medical, gynecologic, or iatrogenic condition (e.g., vulvar surgery) that could explain the presence of chronic vulvar pain (e.g., genitourinary syndrome of menopause, lichen sclerosus, vaginismus, significant pelvic organ prolapse, pudendal neuralgia)
* Active vulvar and/or vaginal infection that is not due to bacterial vaginosis, Chlamydia, Trichomonads or Candida (if diagnosed with any of these infections, treat and re-evaluate after negative test of cure)
* Active urinary tract infection
* Currently pregnant or breastfeeding
* Recent vaginal delivery (within 3 months post-partum)
* Medical or psychiatric condition not under control
* Scoring of 10 or above on the PHQ-9 and/or scoring 1 or above on the question asking about "thoughts that you would be better off dead, or of hurting yourself in some way"
* History of treatment with fractional CO2 laser to the vulvar vestibule and/or vagina
* History of radiation to vaginal/colorectal tissue, reconstructive pelvic surgery with "mesh kits", impaired wound healing or keloid formation, and/or thromboembolic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in subjects' vulvar pain NRS scores | 24 weeks
  The primary outcome will be the mean change from baseline in subjects' vulvar pain NRS scores at 6, 12, 16, and 24 weeks post-randomization. At baseline and at each of these time points, subjects will be asked to rate their vulvar pain in the previous 4 weeks. The question posed to subjects will be worded as follows: "Please indicate, on a scale of 0 to 10, where 0 is no pain at all and 10 is the worst pain you have ever felt, the number that best describes the intensity of your vulvar pain with intercourse, on average, in the past 4 weeks. If intercourse has not been attempted, then indicate the number that best describes the intensity of your vulvar pain with other activities that elicit pain (for example, tampon insertion) in the past 4 weeks." NRS - Numeric Rating Scale - widely used clinically for the assessment of pain. A higher score would represent more pain and a poorer outcome than a lower score.

SECONDARY OUTCOMES:
Mean change from baseline in subjects' scores on pain severity subscale VPAQ | 24 weeks
  The Vulvar Pain Assessment Questionnaire (VPAQ) was developed to assess the dimensions of the pain experience in studies of chronic pain. It consists of 6 primary (pain severity, emotional response, cognitive response, and interference with life, sexual function, and self-stimulation/penetration) and 3 supplementary subscales (pain quality, coping skills, and partner factors). The pain severity subscale of the VPAQ consists of 3 pairs of verbal rating scales (VRS) that test both pain intensity and pain affect (i.e., the emotional response generated by the feeling of pain). Each VRS is a 5-point scale with the following options: none=0, mild=1, moderate=2, severe=3, and worst possible=4, with a mean being calculated to produce the overall score for this subscale. The scale is 0-4 with 4 being the worst possible outcomes.
Mean change from baseline in subjects' scores on pain severity subscale SF-MPQ | 24 weeks
  The Short-Form McGill Pain Questionnaire (SF-MPQ), a well-validated measure of both pain affect and pain quality, consists of 15 pain descriptors rated on a 4-point VRS (none=0, mild=1, moderate=2, severe=3) to yield a total score on a scale from 0-60, where a lower score would represent less pain and a better outcome.
Mean change from baseline in subjects' scores on pain descriptors subscale VPAQ | 24 weeks
  The Vulvar Pain Assessment Questionnaire (VPAQ) was developed to assess the dimensions of the pain experience in studies of chronic pain. It consists of 6 primary (pain severity, emotional response, cognitive response, and interference with life, sexual function, and self-stimulation/penetration) and 3 supplementary subscales (pain quality, coping skills, and partner factors). The pain descriptors subscale of the VPAQ tests pain quality (i.e., how the pain is described in terms of sensory descriptors). It consists of 10 adjectives rated on a 5-point VRS (not at all=0, a little=1, somewhat=2, a lot=3, very much=4) to yield a total score from the mean of the adjectives to represent this subscale. The scale is 0-4 with 4 being the worst outcome.
Mean change from baseline in subjects' scores on the SF-36 | 24 weeks
  The 36-item Short-Form Health Survey (SF-36) consists of 36 questions assessing physical functioning, role functioning difficulties caused by physical problems, bodily pain, general health, vitality, social functioning, role functioning difficulties caused by emotional problems, and mental health. Scoring the SF-36 is a two-step process. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Scale scores represent the average for all items in the scale that the respondent answered. High scores are representative of a great health status and better outcomes, while low scores are representative of a poor health status.
Mean change from baseline in subjects' scores on the pain interference subscale of the BPI | 24 weeks
  The pain interference subscale of the Brief Pain Inventory (BPI), also a generic measure, assesses the degree to which a chronic pain condition interferes with 7 general life domains: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The scale goes from 0-10 with 10 being the worst. It assesses pain at its worst, lease, average, and now (current pain).The mean score for the interference of all of the activities for each severity item (worst, least, average, now) is calculated with a higher score (near 10) being a worse outcome.
Mean change from baseline in subjects' scores on the life interference subscale of the VPAQ | 24 weeks
  The Vulvar Pain Assessment Questionnaire (VPAQ) was developed to assess the dimensions of the pain experience in studies of chronic pain. It consists of 6 primary (pain severity, emotional response, cognitive response, and interference with life, sexual function, and self-stimulation/penetration) and 3 supplementary subscales (pain quality, coping skills, and partner factors). The life interference subscale of the VPAQ tests interference of pain with normal life activities. It consists of 11 everyday activities that could be interrupted by pain rated on a 5-point VRS (not at all=0, a little=1, somewhat=2, a lot=3, very much/I avoid because of pain=4) to yield a total score from the mean of the activities to represent this subscale. The scale is 0-4 with 4 being the worst outcome.
Mean change from baseline in subjects' scores on the life interference subscale of the FSFI | 24 weeks
  The Female Sexual Function Index (FSFI), the most-commonly used generic measure of sexual function in women in PVD studies, consists of 6 subscales related to sexual desire (2 Qs scale 1 worst - 5 best), arousal (4Qs 0 worst - 5 best), lubrication (4Qs 0 worst - 5 best), orgasm (3Qs 0 worst - 5 best), satisfaction (3Qs 0 worst - 5 best), and pain (3Qs 0 worst - 5 best). The sexual function interference subscale of the VPAQ assesses the impact of chronic vulvovaginal pain on sexual function. Higher scores indicate higher sexual functioning, with an overall range of 2-36.. A score of 26.55 has been clinically selected as the cut-off for sexual dysfunction, with a score lower than that indicating this problem.
Mean change from baseline in subjects' scores on the sexual function interference subscale of the VPAQ | 24 weeks
  The Vulvar Pain Assessment Questionnaire (VPAQ) was developed to assess the dimensions of the pain experience in studies of chronic pain. It consists of 6 primary (pain severity, emotional response, cognitive response, and interference with life, sexual function, and self-stimulation/penetration) and 3 supplementary subscales (pain quality, coping skills, and partner factors). The sexual function interference subscale of the VPAQ tests interference of pain with sexual activities. It consists of 10 sexual activities that could be interrupted by pain rated on a 5-point VRS (not at all=0, a little=1, somewhat=2, a lot=3, very much/I avoid because of pain=4) to yield a total score from the mean of the activities to represent this subscale. The scale is 0-4 with 4 being the worst outcome.
Mean change from baseline in subjects' scores on the sexual function interference subscale of the PHQ-9 | 24 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is 1 of 3 scales recommended by the National Institute for Health and Clinical Excellence for use in primary care to measure baseline depression severity and responsiveness to treatment. The scale goes from 0-27 with 0-4 indicating minimal depression with treatment unlikely to be necessary, 5-9 indicating mild depression and 10-14 indicating moderate depression with physicians using their clinical judgement for treatment (score 5-14) based on individual patient, 15-19 indicating moderately severe depression and 20-27 indicating severe depression warrant treatment for the depression (score >14). A higher score would represent a poorer outcome for this scale.
Comparison of percentages of subjects in each treatment arm endorsing improvement in symptoms on the PGIC scale | 24 weeks
  The Patient Global Impression of Change (PGIC) is a 7-point scale that rates the level of satisfaction with treatment (very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse). 10 point scale with 0=much better, 5=no change, and 10=much worse. Scores less than 5 would represent good outcomes. .

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Matthews, MD, Principal Investigator — Professor or Ob/Gyn and Urology
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bornstein J, Goldstein AT, Stockdale CK, Bergeron S, Pukall C, Zolnoun D, Coady D; consensus vulvar pain terminology committee of the International Society for the Study of Vulvovaginal Disease (ISSVD); International Society for the Study of Women's Sexual Health (ISSWSH); International Pelvic Pain Society (IPPS). 2015 ISSVD, ISSWSH, and IPPS Consensus Terminology and Classification of Persistent Vulvar Pain and Vulvodynia. J Sex Med. 2016 Apr;13(4):607-12. doi: 10.1016/j.jsxm.2016.02.167. Epub 2016 Mar 25. PMID 27045260
- [Background] Harlow BL, Kunitz CG, Nguyen RH, Rydell SA, Turner RM, MacLehose RF. Prevalence of symptoms consistent with a diagnosis of vulvodynia: population-based estimates from 2 geographic regions. Am J Obstet Gynecol. 2014 Jan;210(1):40.e1-8. doi: 10.1016/j.ajog.2013.09.033. Epub 2013 Sep 28. PMID 24080300
- [Background] Sadownik LA. Etiology, diagnosis, and clinical management of vulvodynia. Int J Womens Health. 2014 May 2;6:437-49. doi: 10.2147/IJWH.S37660. eCollection 2014. PMID 24833921
- [Background] Falsetta ML, Foster DC, Bonham AD, Phipps RP. A review of the available clinical therapies for vulvodynia management and new data implicating proinflammatory mediators in pain elicitation. BJOG. 2017 Jan;124(2):210-218. doi: 10.1111/1471-0528.14157. Epub 2016 Jun 17. PMID 27312009
- [Background] Salvatore S, Leone Roberti Maggiore U, Athanasiou S, Origoni M, Candiani M, Calligaro A, Zerbinati N. Histological study on the effects of microablative fractional CO2 laser on atrophic vaginal tissue: an ex vivo study. Menopause. 2015 Aug;22(8):845-9. doi: 10.1097/GME.0000000000000401. PMID 25608269
- [Background] Sokol ER, Karram MM. An assessment of the safety and efficacy of a fractional CO2 laser system for the treatment of vulvovaginal atrophy. Menopause. 2016 Oct;23(10):1102-7. doi: 10.1097/GME.0000000000000700. PMID 27404032
- [Background] Pitsouni E, Grigoriadis T, Tsiveleka A, Zacharakis D, Salvatore S, Athanasiou S. Microablative fractional CO2-laser therapy and the genitourinary syndrome of menopause: An observational study. Maturitas. 2016 Dec;94:131-136. doi: 10.1016/j.maturitas.2016.09.012. Epub 2016 Sep 16. PMID 27823733
- [Background] Salvatore S, Nappi RE, Parma M, Chionna R, Lagona F, Zerbinati N, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. Sexual function after fractional microablative CO(2) laser in women with vulvovaginal atrophy. Climacteric. 2015 Apr;18(2):219-25. doi: 10.3109/13697137.2014.975197. Epub 2014 Dec 16. PMID 25333211
- [Background] Zerbinati N, Serati M, Origoni M, Candiani M, Iannitti T, Salvatore S, Marotta F, Calligaro A. Microscopic and ultrastructural modifications of postmenopausal atrophic vaginal mucosa after fractional carbon dioxide laser treatment. Lasers Med Sci. 2015 Jan;30(1):429-36. doi: 10.1007/s10103-014-1677-2. Epub 2014 Nov 20. PMID 25410301
- [Background] Murina F, Karram M, Salvatore S, Felice R. Fractional CO2 Laser Treatment of the Vestibule for Patients with Vestibulodynia and Genitourinary Syndrome of Menopause: A Pilot Study. J Sex Med. 2016 Dec;13(12):1915-1917. doi: 10.1016/j.jsxm.2016.10.006. Epub 2016 Nov 15. PMID 27864031
- [Background] Foster DC, Kotok MB, Huang LS, Watts A, Oakes D, Howard FM, Poleshuck EL, Stodgell CJ, Dworkin RH. Oral desipramine and topical lidocaine for vulvodynia: a randomized controlled trial. Obstet Gynecol. 2010 Sep;116(3):583-593. doi: 10.1097/AOG.0b013e3181e9e0ab. PMID 20733439
- [Background] Gu AP, Gu CN, Ahmed AT, Murad MH, Wang Z, Kallmes DF, Brinjikji W. Sham surgical procedures for pain intervention result in significant improvements in pain: systematic review and meta-analysis. J Clin Epidemiol. 2017 Mar;83:18-23. doi: 10.1016/j.jclinepi.2016.12.010. Epub 2017 Jan 4. PMID 28063914
- [Background] Ciccozzi M, Menga R, Ricci G, Vitali MA, Angeletti S, Sirignano A, Tambone V. Critical review of sham surgery clinical trials: Confounding factors analysis. Ann Med Surg (Lond). 2016 Oct 29;12:21-26. doi: 10.1016/j.amsu.2016.10.007. eCollection 2016 Dec. PMID 27872745
- [Background] Dargie E, Holden RR, Pukall CF. The Vulvar Pain Assessment Questionnaire inventory. Pain. 2016 Dec;157(12):2672-2686. doi: 10.1097/j.pain.0000000000000682. PMID 27780177
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Pukall CF, Bergeron S, Brown C, Bachmann G, Wesselmann U; Vulvodynia Collaborative Research Group. Recommendations for Self-Report Outcome Measures in Vulvodynia Clinical Trials. Clin J Pain. 2017 Aug;33(8):756-765. doi: 10.1097/AJP.0000000000000453. PMID 27841834
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Smarr KL, Keefer AL. Measures of depression and depressive symptoms: Beck Depression Inventory-II (BDI-II), Center for Epidemiologic Studies Depression Scale (CES-D), Geriatric Depression Scale (GDS), Hospital Anxiety and Depression Scale (HADS), and Patient Health Questionnaire-9 (PHQ-9). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S454-66. doi: 10.1002/acr.20556. No abstract available. PMID 22588766
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Schreiber, J., Culpeper, L. Suicidal ideation and behavior in adults. In: UpToDate, Post TW (Ed), UpToDate, Waltham, MA. (Accessed on June 13, 2017.)
- [Background] Bergeron S, Khalife S, Dupuis MJ, McDuff P. A randomized clinical trial comparing group cognitive-behavioral therapy and a topical steroid for women with dyspareunia. J Consult Clin Psychol. 2016 Mar;84(3):259-68. doi: 10.1037/ccp0000072. Epub 2016 Jan 4. PMID 26727408
- [Background] Bergeron S, Binik YM, Khalife S, Pagidas K, Glazer HI, Meana M, Amsel R. A randomized comparison of group cognitive--behavioral therapy, surface electromyographic biofeedback, and vestibulectomy in the treatment of dyspareunia resulting from vulvar vestibulitis. Pain. 2001 Apr;91(3):297-306. doi: 10.1016/S0304-3959(00)00449-8. PMID 11275387
- [Background] Fitzmaurice GM, Ravichandran C. A primer in longitudinal data analysis. Circulation. 2008 Nov 4;118(19):2005-10. doi: 10.1161/CIRCULATIONAHA.107.714618. No abstract available. PMID 18981315